CLINICAL TRIAL: NCT03755947
Title: Sequential Triple Therapy With Ibrutinib, Obinutuzumab and Venetoclax in First and Second Line for Patients With Chronic Lymphocytic Leukemia
Brief Title: Ibrutinib, Obinutuzumab and Venetoclax for Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Cooperativo de Hemopatías Malignas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAL 306/2018
Record Dates: First submitted 2018-11-20; First posted 2018-11-28 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: B-Cell Chronic Lymphocytic Leukemia; B-Cell Chronic Lymphocytic Leukemia in Relapse (Diagnosis)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Disease | interventions — ibrutinib; obinutuzumab; venetoclax

STUDY DESIGN:
Intervention Model Description: This is a multicenter, longitudinal, experimental, open, non-randomized and non-comparable study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IGV (Experimental): Cytoreduction 3 cycles (I) Ibrutinib, [Imbruvica, Janssen]
  Induction 6 cycles (G) Obinutuzumab, [Gazyva, Roche]
  Consolidation 12 cycles (V) Venetoclax, [Venclexta, Abbvie].
  Interventions: Drug: Ibrutinib; Drug: Obinutuzumab; Drug: Venetoclax

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib Oral Capsule [Imbruvica] Tablets 120 mg. Oral. 420mg/day, day 1 to 28, every 28 days. 3 cycles.
  Other Names: Imbruvica
Drug: Obinutuzumab — Obinutuzumab Injection. Intravenous Solution [Gazyva] Parenteral. 1000 mg, day 1 of every cycle, every 28 days. 6 cycles.
  Other Names: Gazyva
Drug: Venetoclax — Venetoclax Oral Tablets [Venclexta] Tablets 100 mg. Oral. 400 mg/day. Day 1 to 28, every 28 days. 12 cycles.
  Other Names: Venclexta

SUMMARY:
Background: Chronic Lymphocytic Leukemia (CLL) is the most common leukemia in the occidental countries. Until now, it is considered a chronic disease without a cure. The development of new molecular therapies have showed that the cure may be an option. This protocol propose a triple sequential therapy with three direct therapies for the leukemic cell: an inhibitor of Bruton´s tyrosine kinase (ibrutinib), a second generation monoclonal antibody versus CD20 (obinutuzumab) and a BCL-2 inhibitor (venetoclax) as treatment of first or second line in CLL.

Objective: Negativize the minimal residual disease and by this way obtain longer survivals (overall survival and relapse free survival).

Design: This is a multicenter, longitudinal, experimental, open, non-randomized and non-comparable study coordinated by the "Grupo Cooperativo de Hemopatías Malignas" situated on Hospital Angeles Lomas in Huixquilucan, México. The study, is a phase II clinical study that will employ three target therapy drugs in sequencing phases. It will start with a BTK inhibitor as induction, later an anti-CD20 will be used for consolidation and it will end with a BH3 analog as maintenance for one year. The primary outcome is the negativization of minimal residual disease.

DETAILED DESCRIPTION:
The international recommendations indicate that the first line of treatment for patients <65 years old and with no significant comorbidities (fit patients) the known regime of FCR with recommendation of category 1 and later bendamustine with antiCD20 or ibrutinib. For patients >65 years old or not fit for intensive treatment it is recommended chlorambucil with obinutuzumab, monotherapy with ibrutinib, bendamustine with antiCD20 or chlorambucil with another antiCD20 like rituximab or ofatumumab. In case of patients with high-risk alterations of relapse due to positive MRD at the end of the treatment it is recommended a maintenance schedule with lenalidomide.

The antibodies against CD20 have shown through the years its activity in diverse alterations of B-cells. Rituximab was approved in 1998 for B-cells Non-Hodgkin lymphomas including CLL. Currently there are new anti-CD20 with more activity than rituximab. One of them is obinutuzumab which, by the monoclonal antibody engineering shows a greater affinity to the union of the epitope CD20 generating increased cellular cytotoxicity.

Bruton's tyrosine kinase (BTK), generates signaling cascades for the cell survival by the NF-KB and MAP kinases way, which leads to the transduction of the B cell receptor (BCR). Ibrutinib is a molecule that inhibits BTK inducing apoptosis in the B cells being currently used in the diverse mature B cell neoplasms.

Another therapeutic target is the BCL-2 protein (B-cell lymphoma 2) which is a key regulator in the apoptotic and it's compromised in the B cell neoplasms. Venetoclax is a mimetic drug to BH3 that blocks the function of BCL-2.

Based in the old and new drugs described in CLL, there is a great number of combinations that can be applied in the different phases of the disease as well as by risk stages and physical state of the patient. Before this scenario diverse CLL study groups proposes the strategy of sequencing in three phases (triple T) trying to prevent the development of leukemic subclones, minimize the use of chemotherapy that generates secondary mutations in CLL and other neoplasms. These type of treatment counts with the advantage of: 1) being available for patients physically fit or not due to the a limited toxicity of the drugs, 2) applying in an out-of-hospital environment and 3) adjusting the treatment according to the response to generate an effective cost in the new drugs. Thus, it is proposed the cytoreduction sequencing for 1 to 2 cycles, induction for 6 to 12 months and the MRD maintenance that could go from one year up to undefined with ibrutinib, obinutuzumab and venetoclax in that order.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with B cell chronic lymphocytic leukemia according to 2017 WHO criteria by immunophenotype/immunohistochemistry with active disease according to the 2018 International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria and do not present TP53 mutation and/or del(17)p. (Cohort 1).
* Patients diagnosed with relapsed/refractory chronic lymphocytic leukemia that have previously received at least one line of treatment that does not include the drugs in the study scheme. (Cohort 2).
* Functional stage of 0 - 2 measured by the Eastern Cooperative Oncology Group (ECOG) scale.
* Creatinine depuration ≥ 30 ml/min measured in a 24-hour urine recollection or utilizing the CKD-EPI formula.
* Proper liver function: total bilirubin ≤ 1.5 x upper limit of normal (ULN) or ≤ 3 x ULN in patients with Gilbert syndrome, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 x ULN.
* Capacity and willingness to provide a written informed consent.

Exclusion Criteria:

* T cell lymphocytic leukemia diagnosis.
* TP53 mutation and/or del(17)p presence.
* Non-controlled systematic active infection (viral, bacterial and/or fungic).
* Patients with known infection by human immunodeficiency virus (HIV).
* Active infection by hepatitis B (defined as the presence of detectable HBV's DNA, HBe antigen or HBs antigen). Patients with serological evidence of previous vaccination (HBsAg negative, anti-HBs positive antibodies, anti-HBc negative antibodies) are eligible. The patients that are HBsAg negative/ anti-Hbs positive antibodies but anti-HBc positive antibodies are eligible, if the HBV DNA is negative, and the HBV-DNA PCR is realized every 12 months after the last cycle of treatment.
* Active infection by hepatitis C, defined by the ribonucleic acid (RNA) of hepatitis C is detectable in plasma by polymerase chain reaction (PCR).
* Significant cardiovascular diseases such as uncontrolled or symptomatic arrhythmias, congestive heart failure or acute myocardial infarction within 2 months prior to screening, or any class 3 or 4 heart disease according to the functional classification of the NYHA.
* Diagnosis of previous malignancies for 2 years, with exception of patients with basal or squamous cell carcinoma or "in situ" carcinoma of cervix or breast.
* Requiring therapy with inhibitors or potent inducers of CYP3A4 and CYP3A5 inhibitors.
* Anticoagulant therapy with acenocoumarol or warfarin.
* History of cerebrovascular accident or intracranial hemorrhage within 6 months prior to screening.
* History of allergic reaction or severe anaphylaxis to humanized or murine monoclonal antibodies.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Best response obtained | Two months after finishing the triple sequencing therapy
  The best response obtained will be defined as CR with negative MRD by the iwCLL response criteria measured subsequent a cytoreduction treatment, induction and consolidation with the triple sequencing therapy with Ibrutinib, Obinutuzumab and Venetoclax in patients with chronic lymphocytic leukemia.

SECONDARY OUTCOMES:
Overall Survival | Three years
  Defined as the time since the end of treatment to time of death in the patients diagnosed with chronic lymphocytic leukemia in treatment with a triple sequencing therapy with Ibrutinib, Obinutuzumab and Venetoclax
Relapse-Free Survival | Three years
  Defined as the time since the end of treatment to time to relapse in the patients diagnosed with chronic lymphocytic leukemia in treatment with a triple sequencing therapy with Ibrutinib, Obinutuzumab and Venetoclax
Rate of AcuteToxicity | Two years
  Adverse effects associated to triple sequencing therapy with Ibrutinib, Obinutuzumab and Venetoclax
Rate of Late Toxicity | Three years
  Adverse effects associated to triple sequencing therapy with Ibrutinib, Obinutuzumab and Venetoclax on long term follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo Cooperativo de Hemopatías Malignas, Huixquilucan, State of Mexico, Mexico

REFERENCES:
- [Background] Hallek M, Cheson BD, Catovsky D, Caligaris-Cappio F, Dighiero G, Dohner H, Hillmen P, Keating M, Montserrat E, Chiorazzi N, Stilgenbauer S, Rai KR, Byrd JC, Eichhorst B, O'Brien S, Robak T, Seymour JF, Kipps TJ. iwCLL guidelines for diagnosis, indications for treatment, response assessment, and supportive management of CLL. Blood. 2018 Jun 21;131(25):2745-2760. doi: 10.1182/blood-2017-09-806398. Epub 2018 Mar 14. PMID 29540348
- [Background] Rai KR, Jain P. Chronic lymphocytic leukemia (CLL)-Then and now. Am J Hematol. 2016 Mar;91(3):330-40. doi: 10.1002/ajh.24282. PMID 26690614
- [Background] Garcia Marco JA, Giraldo Castellano P, Lopez Jimenez J, Rios Herranz E, Sastre Moral JL, Terol Castera MJ, Bosch Albareda F; en representacion del Grupo Espanol de Leucemia Linfatica Cronica (GELLC); Sociedad Espan ola de Hematologi a y Hemoterapia. [National guidelines for the management of patients with chronic lymphocytic leukemia. Sociedad Espan ola de Hematologi a y Hemoterapia and Grupo Espan ol de Leucemia Linfoci tica Cro nica]. Med Clin (Barc). 2013 Aug 17;141(4):175.e1-8. doi: 10.1016/j.medcli.2013.04.041. Epub 2013 Jul 3. Spanish. PMID 23830547
- [Background] Cartron G, de Guibert S, Dilhuydy MS, Morschhauser F, Leblond V, Dupuis J, Mahe B, Bouabdallah R, Lei G, Wenger M, Wassner-Fritsch E, Hallek M. Obinutuzumab (GA101) in relapsed/refractory chronic lymphocytic leukemia: final data from the phase 1/2 GAUGUIN study. Blood. 2014 Oct 2;124(14):2196-202. doi: 10.1182/blood-2014-07-586610. Epub 2014 Aug 20. PMID 25143487
- [Background] Farooqui MZ, Valdez J, Martyr S, Aue G, Saba N, Niemann CU, Herman SE, Tian X, Marti G, Soto S, Hughes TE, Jones J, Lipsky A, Pittaluga S, Stetler-Stevenson M, Yuan C, Lee YS, Pedersen LB, Geisler CH, Calvo KR, Arthur DC, Maric I, Childs R, Young NS, Wiestner A. Ibrutinib for previously untreated and relapsed or refractory chronic lymphocytic leukaemia with TP53 aberrations: a phase 2, single-arm trial. Lancet Oncol. 2015 Feb;16(2):169-76. doi: 10.1016/S1470-2045(14)71182-9. Epub 2014 Dec 31. PMID 25555420
- [Background] Byrd JC, Brown JR, O'Brien S, Barrientos JC, Kay NE, Reddy NM, Coutre S, Tam CS, Mulligan SP, Jaeger U, Devereux S, Barr PM, Furman RR, Kipps TJ, Cymbalista F, Pocock C, Thornton P, Caligaris-Cappio F, Robak T, Delgado J, Schuster SJ, Montillo M, Schuh A, de Vos S, Gill D, Bloor A, Dearden C, Moreno C, Jones JJ, Chu AD, Fardis M, McGreivy J, Clow F, James DF, Hillmen P; RESONATE Investigators. Ibrutinib versus ofatumumab in previously treated chronic lymphoid leukemia. N Engl J Med. 2014 Jul 17;371(3):213-23. doi: 10.1056/NEJMoa1400376. Epub 2014 May 31. PMID 24881631
- [Background] Barr PM, Robak T, Owen C, Tedeschi A, Bairey O, Bartlett NL, Burger JA, Hillmen P, Coutre S, Devereux S, Grosicki S, McCarthy H, Li J, Simpson D, Offner F, Moreno C, Zhou C, Styles L, James D, Kipps TJ, Ghia P. Sustained efficacy and detailed clinical follow-up of first-line ibrutinib treatment in older patients with chronic lymphocytic leukemia: extended phase 3 results from RESONATE-2. Haematologica. 2018 Sep;103(9):1502-1510. doi: 10.3324/haematol.2018.192328. Epub 2018 Jun 7. PMID 29880603
- [Background] Roberts AW, Davids MS, Pagel JM, Kahl BS, Puvvada SD, Gerecitano JF, Kipps TJ, Anderson MA, Brown JR, Gressick L, Wong S, Dunbar M, Zhu M, Desai MB, Cerri E, Heitner Enschede S, Humerickhouse RA, Wierda WG, Seymour JF. Targeting BCL2 with Venetoclax in Relapsed Chronic Lymphocytic Leukemia. N Engl J Med. 2016 Jan 28;374(4):311-22. doi: 10.1056/NEJMoa1513257. Epub 2015 Dec 6. PMID 26639348
- [Background] Cramer P, von Tresckow J, Bahlo J, Robrecht S, Langerbeins P, Al-Sawaf O, Engelke A, Fink AM, Fischer K, Tausch E, Seiler T, Fischer von Weikersthal L, Hebart H, Kreuzer KA, Bottcher S, Ritgen M, Kneba M, Wendtner CM, Stilgenbauer S, Eichhorst B, Hallek M. Bendamustine followed by obinutuzumab and venetoclax in chronic lymphocytic leukaemia (CLL2-BAG): primary endpoint analysis of a multicentre, open-label, phase 2 trial. Lancet Oncol. 2018 Sep;19(9):1215-1228. doi: 10.1016/S1470-2045(18)30414-5. Epub 2018 Aug 13. PMID 30115596
- [Background] Fischer K, Al-Sawaf O, Fink A-M, et al. Venetoclax and obinutuzumab in chronic lymphocytic leukemia. Blood. 2017;129(19):2702-2705. Blood. 2017 Jul 13;130(2):232. doi: 10.1182/blood-2017-05-787366. No abstract available. PMID 28705863
- [Background] Seymour JF, Kipps TJ, Eichhorst B, Hillmen P, D'Rozario J, Assouline S, Owen C, Gerecitano J, Robak T, De la Serna J, Jaeger U, Cartron G, Montillo M, Humerickhouse R, Punnoose EA, Li Y, Boyer M, Humphrey K, Mobasher M, Kater AP. Venetoclax-Rituximab in Relapsed or Refractory Chronic Lymphocytic Leukemia. N Engl J Med. 2018 Mar 22;378(12):1107-1120. doi: 10.1056/NEJMoa1713976. PMID 29562156
- [Background] Hallek M. Signaling the end of chronic lymphocytic leukemia: new frontline treatment strategies. Blood. 2013 Nov 28;122(23):3723-34. doi: 10.1182/blood-2013-05-498287. Epub 2013 Sep 24. PMID 24065239